CLINICAL TRIAL: NCT00814034
Title: An Observational, Prospective Cohort Study, on Blood Coagulation Parameters in Postmenopausal Patients With Operable Breast Cancer Who Are Treated as Per Standard Practice With Adjuvant Hormonal Therapy for a Total of 5 Years
Brief Title: Coagulation Parameters in Postmenopausal Breast Cancer Patients Under Adjuvant Hormonal Therapy
Acronym: COPA
Status: Completed | Type: Observational
Sponsor: Hellenic Breast Surgeons Society (Other)
Responsible Party: Principal Investigator, Markopoulos Christos, Professor of Surgery, Athens University Medical School, Hellenic Breast Surgeons Society
Other Study IDs: COPA-HBSS0801
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: Aromatase Inhibitors; Coagulation parameters; Tamoxifen
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1:Tamoxifen
- 2:Steroidal Aromatase Inhibitor
- 3:Non-steroidal Aromatase Inhibitor

SUMMARY:
The objective of the study is to monitor the changes of blood coagulation parameters in postmenopausal patients who are treated with adjuvant Hormonal Therapy for a total of 5 years. The values of the standard coagulation parameters throughout the study will be compared with the baseline values.

DETAILED DESCRIPTION:
Study subjects will be treated with standard adjuvant hormonal therapy for a total of 5 years or until disease relapse or until HT is permanently discontinued for other reasons. The choice of endocrine treatment strategy (drugs to be used or their sequence, if the sequential option has been decided) is left at the discretion of the participating site. Adjuvant HT will commence after the completion of adjuvant chemotherapy and/or radiotherapy. Percentage change (%) from baseline of the blood coagulation parameters at 6, 12, 18, and 24 months of treatment. The blood coagulation parameters which will be measured are fibrinogen, prothrombin time (PT) and activated partial thromboplastin time (aPTT).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status. ER and/or PgR status positive. Adjuvant hormonal treatment for 5 years according to standard practice has been decided by the treating physician. Values within normal limits for the blood coagulation parameters at baseline visit. Accessible for follow-up for the duration of the trial. Written informed consent.

Exclusion Criteria:

* Both ER and PgR negative primary tumor. Evidence of distant metastases (M1) Neo-adjuvant hormonotherapy. Chronic use of oral anticoagulants such as warfarin or acenocoumarol. Psychiatric disorders preventing proper informed consent. Concomitant malignancies except for adequately treated carcinoma in situ of the uterine cervix or basal squamous cell carcinoma of the skin.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal, ER and/or PgR positive breast cancer patients eligible for adjuvant hormonal treatment (HT), who are admitted for treatment and follow-up at the participating sites, will be enrolled in the trial. Study subjects will be treated with standard adjuvant hormonal therapy for a total of 5 years or until disease relapse or until HT is permanently discontinued for other reasons.
  The choice of endocrine treatment strategy (drugs to be used or their sequence, if the sequential option has been decided) is left at the discretion of the participating site. Adjuvant HT will commence after the completion of adjuvant chemotherapy and/or radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage change (%) from baseline of the blood coagulation parameters (fibrinogen, PT, aPTT) at 6, 12, 18, and 24 months of treatment. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christos Markopoulos, MD, Principal Investigator — Hellenic Breast Surgeons Society
Locations (2):
- Greece (2):
  - Hellenic Breast Surgeons Society, Athens, Attica
  - Hellenic Breast Surgeons Society, Athens